CLINICAL TRIAL: NCT01014572
Title: The Effect of Exercise and Alagebrium on the Diastolic Function of the Heart
Acronym: AGE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Benjamin Levine, Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STU 122010-189; R01AG017479 (NIH); IRB#032008-012; IND72,382
Record Dates: First submitted 2009-11-13; First posted 2009-11-17 (Estimated); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Ventricular Function
Keywords: Clinical Trials, Phase II; Exercise; Exercise Tolerance; Aging
MeSH Terms: conditions — Motor Activity | interventions — alagebrium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Aerobic Exercise Training + Placebo (Experimental)
  Interventions: Behavioral: Aerobic Exercise Training
- Tai Chi and/or Yoga Training + Placebo (Experimental)
  Interventions: Behavioral: Tai Chi and/or Yoga Training
- Aerobic Exercise Training + Alagebrium (Experimental)
  Interventions: Behavioral: Aerobic Exercise Training; Drug: Alagebrium (generic: ALT-711)
- Tai Chi and/or Yoga Training + Alagebrium (Experimental)
  Interventions: Drug: Alagebrium (generic: ALT-711); Behavioral: Tai Chi and/or Yoga Training

INTERVENTIONS:
Behavioral: Aerobic Exercise Training — Aerobic exercise training consisting of exercise of choice (walking, eliptical machine, stairstepper, stationary bike, etc.) 4 times per week for 40 minutes at a base pace, and two higher intensity steady state sessions per month.
  Arms: Aerobic Exercise Training + Alagebrium; Aerobic Exercise Training + Placebo
Drug: Alagebrium (generic: ALT-711) — The dosage of our drug, ALT-711, will be one 100 mg caplet by mouth twice per day for 12 months. Total dose per day 200 mg.
  Arms: Aerobic Exercise Training + Alagebrium; Tai Chi and/or Yoga Training + Alagebrium
Behavioral: Tai Chi and/or Yoga Training — Tai Chi or Yoga training includes a series of exercises that improve flexibility, balance and coordination. Training will be supervised by trained instructors. This training will occur 3 times per week.
  Arms: Tai Chi and/or Yoga Training + Alagebrium; Tai Chi and/or Yoga Training + Placebo

SUMMARY:
The purpose of this study is to determine whether an investigational drug (Alagebrium (generic: ALT-711), a type of medication referred to as an advanced glycaton end-product clever) can be combined with exercise training to reverse the stiffening of the heart that takes place naturally with aging.

DETAILED DESCRIPTION:
Objectives: Chronic physical inactivity contributes to the deaths of nearly 1 in 10 Americans. In seniors, the single most common life-threatening disease is congestive heart failure and for these patients, abnormalities of diastolic function play a critical role in the pathophysiology of their disease. The sponsor's research has demonstrated that healthy but sedentary aging leads to atrophy and stiffening of the heart with reduced myocardial and chamber compliance. In contrast, highly competitive senior runners had cardiac compliance that was indistinguishable from healthy young individuals suggesting that lifelong exercise training prevented this stiffening. However, prolonged and intense exercise training (4-6 hrs/wk for 1 yr) failed to restore cardiac compliance in healthy seniors despite other health benefits.

Why did this year of training fail to restore cardiac compliance? New evidence suggests that the structural plasticity of myocardial cells in the elderly may be functionally constrained by the accumulation of toxic metabolites called advanced glycation end-products (AGEs). AGEs are arrays of protein which have been non-enzymatically cross-linked by sugars; these arrays increase the stiffness of arterial walls and the myocardium. Investigators have recently developed a drug capable of cleaving AGE cross-links. Termed ALT-711, this drug has been shown to be safe in human studies with varying degrees of efficacy on endpoints such as blood pressure and non-invasive indices of diastolic function. Based on animal studies, we hypothesize that AGE cross-links must be broken before a meaningful improvement in cardiac compliance can occur with exercise training in sedentary seniors.

Hypothesis: We hypothesize that AGE cross-links must be broken before a meaningful improvement in cardiac compliance can occur with exercise training in previously sedentary seniors; the combination of the AGE cross-link breaker, ALT-711, with exercise training will be superior to either intervention alone in improving cardiac compliance in these subjects.

Specific Aim: To test this hypothesis, we will study four groups of previously sedentary senior subjects for one year with the following interventions: A) sedentary controls taking placebo; B) sedentary subjects taking ALT-711; C) subjects undergoing moderate intensity exercise training while taking placebo and D) subjects undergoing moderate intensity exercise training while taking ALT-711.

A comprehensive set of "Baseline Testing" (prior to the one year intervention) and "Follow-up Testing" (after the one year intervention) will take place to assess the effects of the intervention. This testing will include submaximal and maximal exercise testing as well as comprehensive invasive (right heart catheterization) and non-invasive (ultrasound, MRI) measures of cardiac mechanics, relaxation and morphology. From these data, the following indices of diastolic and systolic function will be generated: Starling and pressure/volume curves; calculations of LV wall stress and strain; and measurements of flow propagation velocity, ejection fraction and relaxation velocity.

In assessing the risk benefit ratio for our study, the major benefits include: 1) obtaining meaningful information for society regarding the effects of ALT-711 and moderate intensity exercise training on the compliance of the left ventricular chamber; 2) obtaining important information for the subject regarding ambulatory blood pressure, exercise performance, cardiac morphology and cardiac function; and 3) providing the subject one year of supervised moderate intensity exercise training or yoga training, each with associated health benefits. The risks of the study are primarily imposed by the dosing of our investigational drug, which has a favorable side effect profile, and the placement of a peripherally inserted right heart catheter, which carries minimal risk when placed by an experienced cardiovascular specialist in a catheterization lab. Hence, in the final analysis, we feel the benefits to both the enrolled individual and to society far outweigh the risks of participation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy senior status (age > 64)
* Body mass index < 30
* Sedentary status (not exercising > 2/wk)

Exclusion Criteria:

* Hypertension
* Diabetes
* Heart Failure
* Asthma
* Chronic obstructive pulmonary disease
* Coronary artery disease (as evidenced by angina or prior myocardial infarction)
* Cerebrovascular disease (as evidenced by prior transient ischemic attack or stroke)

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 62 (Actual)
Dates: Start 2008-07; Primary Completion 2012-06 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Left ventricular compliance and distensibility. | One year after enrollment in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin D Levine, M.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- The Institute for Exercise and Environmental Medicine, Dallas, Texas, United States

REFERENCES:
- [Derived] Fujimoto N, Hastings JL, Carrick-Ranson G, Shafer KM, Shibata S, Bhella PS, Abdullah SM, Barkley KW, Adams-Huet B, Boyd KN, Livingston SA, Palmer D, Levine BD. Cardiovascular effects of 1 year of alagebrium and endurance exercise training in healthy older individuals. Circ Heart Fail. 2013 Nov;6(6):1155-64. doi: 10.1161/CIRCHEARTFAILURE.113.000440. Epub 2013 Oct 15. PMID 24130005